CLINICAL TRIAL: NCT06978413
Title: Telerehabilitation With Digital Technologies for the Continuum of Care of Stroke Patients: a Multicentre Randomized Controlled Trial on Effectiveness, Acceptability, Usability, and Economic Sustainability
Brief Title: Telerehabilitation With Digital Technologies for the Continuum of Care of Stroke Patients
Acronym: StrokeHomeFit4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Ospedale Policlinico San Martino (Other); C.O.T. Cure Ortopediche Traumatologiche S.p.A. (Other); Università di Pavia (Unknown); Scuola Superiore Sant'Anna di Pisa (Other); Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fit4MedRobStroke@Home; PNC0000007 (Other Grant/Funding Number: Ministry of University and Research of Italy)
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: rehabilitation; telerehabilitation; digital technologies; home-based
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Digital Tools (Experimental): The experimental treatment involves home-based telerehabilitation protocols utilizing digital tools. Patients will perform task-oriented activities aimed at improving balance through standing and/or seated exercises under both static and dynamic conditions. Exercise complexity will be progressively adapted and personalized based on the patient's performance, improvement trajectory, and instrumental feedback from the digital system.
  All devices must have a CE mark for medical devices and be used according to the manufacturer's specifications.
  Interventions: Other: Integrated Treatment with Digital Tools
- Educational Program (Active Comparator): Patients in the Control Group will follow a self-guided educational program supported by printed materials outlining daily living activities to be performed at home.
  Interventions: Other: Home-Based Educational Program

INTERVENTIONS:
Other: Integrated Treatment with Digital Tools — Patients will undergo a 6-week remote telerehabilitation program. The recommended frequency of treatment is a minimum of 3 sessions per week, but patients may adjust the schedule in agreement with their assigned therapist. If a patient is unable to complete at least 18 sessions due to clinical reasons, they will be considered as a dropout.
  Moreover, one session per week will be conducted synchronously, with the therapist remotely supervising the patient's activities in real time, while the remaining sessions will be asynchronous, allowing the patient to complete the exercises independently.
  Arms: Treatment with Digital Tools
Other: Home-Based Educational Program — Patients will be monitored over a six-week period through weekly phone calls to assess their progress and overall condition. Additionally, participants are required to maintain an activity diary to document their engagement with the prescribed activities.
  Arms: Educational Program

SUMMARY:
The goal of the pragmatic study is to evaluate the effectiveness of a home-based telerehabilitation protocol for patients with post-stroke disabilities, compared to a home-based educational program.

The main question it aims to answer is:

Is home-based neuromotor and cognitive rehabilitation using digital tools more effective than a traditional educational program for improving static and dynamic balance in patients with subacute and chronic stroke? Researchers will compare the outcome (Berg Balance Scale) measured at baseline with the outcome after treatment to test its effectiveness.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of a home-based treatment based on rehabilitation technologies by comparing it with a traditional educational program at home.

Primary objective: Demonstration of the superiority of a home-based rehabilitation program with digital tools (home-based technological telerehabilitation) over a home-based educational program (home-based usual care) in patients with stroke outcomes in improving static and dynamic balance.

Secondary objectives:

* Evaluation of the impact of the frequency of the intervention on recovery;
* Evaluation of the acceptability of the intervention with digital tools for the patient, the caregiver, and the health care provider;
* Evaluation of the usability of the intervention with digital tools for the patient and the caregiver;
* Evaluation of the economic sustainability of the integrated rehabilitation intervention with digital tools for the patient, the payer, and society through the creation of a cost-effectiveness, cost-utility, and, for the health system, budget impact analysis model evaluation and prediction, and related sensitivity analyses.

The study is designed as a multicenter, multimodal, randomized, controlled, parallel group (1:1), blinded interventional trial. It will be conducted at multiple clinical centers participating in a national research initiative. Randomization will be centralized and stratified by clinical center, time since stroke, and age.

The sample size was determined using a 2-tailed, 2-sample t-test, assuming a power of 80%, a type I error t of 0.05, a mean difference of 2.7 units on the primary outcome (specifically, the change in the Berg Balance Scale, corresponding to the minimum detectable change in chronic stroke patients) and a common standard deviation of 5.37 points. With these assumptions, a sample size of 128 cases was estimated. Further, considering a dropout rate of 20%, the final estimated sample size required is 160 cases. The calculation was performed using G*Power software.

All participating centers will follow a standardized operating procedure regarding treatment and outcome assessment to ensure consistency across all sites. Data will be systematically collected using the REDCap (Research Electronic Data Capture) platform.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of first ischemic or hemorrhagic stroke verified by Computed Axial Tomography or MRI.
* Age greater than 18 years.
* Latency since the event: a) greater than 3 months and less than or equal to 6 months; b) greater than 6 months and less than 24 months.
* Ability to perform the Timed Up and Go Test.

Exclusion Criteria:

* Unstable clinical conditions.
* Behavioral/cognitive disorders that prevent adequate patient compliance with the study (severe cognitive impairment, Montreal Cognitive Assessment<17.5).
* Severe visual impairment that cannot be corrected by lenses, preventing the patient from performing treatment with digital instruments.
* Refusal to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Berg Balance Scale (BBS) | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for the upper extremities - motor function | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The upper extremity motor function domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, and hand. It ranges from 0 (hemiplegia) to 66 (normal motor performance).
Fugl-Meyer Assessment for the upper extremities - sensory function | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The upper extremity sensory function domain evaluates light touch on two surfaces of the arm, and position sense for upper limb joints. It ranges from 0 to 12 (normal sensory function).
Fugl-Meyer Assessment for the lower extremities - motor function | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The lower extremity motor function domain includes items assessing movement, coordination, and reflex action of the hip, knee, and ankle. It ranges from 0 (hemiplegia) to 34 (normal motor performance).
Fugl-Meyer Assessment for the lower extremities - sensory function | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The lower extremity sensory function domain evaluates light touch on two surfaces of the leg, and position sense for lower limb joints. It ranges from 0 to 12 (normal sensory function).
Modified Rivermead Motricity Index | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Modified Rivermead Motricity Index (MRMI) is a clinical tool used to assess motor function and mobility in patients with neurological impairments. It consists of 8 items that evaluate motor control, balance, and mobility, with a total possible score of 40 points. Each item is scored on a 5-point ordinal scale (0-5), with higher scores indicating better function.
Symbol Digit Modalities Test | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Symbol Digit Modalities Test evaluates information processing speed. It consists of a simple task of replacing symbols with numbers. Using a reference key, the patient has 90 seconds to match a sequence of symbols with the correspondent numbers as rapidly as possible. Both written or oral administration can be used. For each correct answer, a point is assigned. The higher the score, the faster the information processing speed.
Modified Barthel Index | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The modified Barthel Index for Activities of Daily Living is a validated ordinal scale which measures a person's ability to complete activities of daily living (ADL). Scores range from 0 (total dependence) to 100 (total independence).
Modified Ashworth Scale | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Modified Ashworth Scale (MAS) is a revised version of the original Ashworth Scale that measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0 to 4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch. The lower the score, the lower the spasticity. Upper and lower joints spasticity is assessed.
Motricity Index for upper extremities | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Motricity Index (MI) is an ordinal method of measuring limb strength. For upper extremity test, shoulder abduction, elbow flexion, pinch grip are considered. It ranges from 0 (worse) to 100 (normal strength).
Motricity Index for lower extremities | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Motricity Index (MI) is an ordinal method of measuring limb strength. For lower extremity test, hip flexion, knee extension, and ankle dorsiflexion are considered. It ranges from 0 (worse) to 100 (normal strength).
Trunk control test | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Trunk control test (TCT) measures four simple aspects of trunk movement. Total score range from 0 (minimum) to 100 (maximum, indicating better performance).
Numerical Rating Scale for Pain | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Numerical Rating Scale fo Pain (NRSP) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Neuropathic Pain 4 Questions | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Neuropathic Pain 4 Questions (DN4) is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Functional Ambulation Classification Scale | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Functional Ambulation Classification (FAC) Scale is a simple and widely used tool to assess a person's ability to walk (ambulate) independently after a neurological injury. It evaluates how much physical support a person needs while walking and helps clinicians classify their functional mobility. The FAC consists of six levels (0-5), ranging from non-functional ambulation to independent walking.
Frontal Assessment Battery | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The Frontal Assessment Battery (FAB) is a clinical tool designed to assess frontal lobe functions, particularly executive functions, which are cognitive processes like problem-solving, decision-making, and impulse control. The FAB consists of six subtests, each scored from 0 to 3, with a maximum total score of 18 points. Higher scores indicate better frontal lobe function.
World Health Organization disability assessment schedule 2.0 - WHODAS 2.0 | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  WHODAS 2.0 assesses the functioning and disability level in six domains (cognition, mobility, self-care, getting along, life activities, and participation in community activities) according to the International Classification of Functioning, Disability and Health (ICF). The summary scores for the WHODAS 2.0 will be obtained through 3 steps: 1) summing of item scores within each domain; 2) summing all six domain scores; 3) converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability and 100 = full disability).
5-level EQ-5D version (EQ-5D-5L) | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  The 5-level EQ-5D version (EQ-5D-5L) is a validated tool to assess health-related quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Index scores range from -0.59 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.

OTHER OUTCOMES:
premorbid Modified Rankin Scale | Baseline
  The pre-stroke Modified Rankin Score (mRS) is an estimated score used to assess the patient's pre-stroke level of function. It has a grade ranging from 0 (no symptoms) to 6 (dead).
Montreal Cognitive Assessment Scale | Baseline
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. It ranges from 0 (worst) to 30 (best).
Timed Up and Go | Baseline
  The Timed Up and Go (TUG) test is a simple and widely used assessment to evaluate mobility, balance, walking ability, and fall risk.The test measures the time (in seconds) it takes for a person to: (i) Stand up from a standard chair (seat height ~46 cm); (ii) Walk 3 meters (10 feet) forward at a comfortable pace; (iii) Turn around at the 3-meter mark; (iv) Walk back to the chair; (v) Sit down again. The total time taken is recorded, with specific cut-off values indicating different levels of mobility impairment and fall risk.
Computer skills questionnaire | Baseline
  It is an ad-hoc questionnaire to assess computer skills. It collects information regarding personal competencies in the use of technology, with items rated on a 5-point scale (1 to 5) to evaluate both the level of knowledge and the frequency of technology use. The questionnaire also includes general information questions about computer skills, assessed using a dichotomous (yes/no) scale.
Technology Acceptance Model | Within 7 days after the end of the 6-week observation/rehabilitation period
  It is a questionnaire used with the primary aim of identifying the determinants involved in the acceptance of Robotic and Allied Technology. The questionnaire consists of 4 sections (perceived usefulness, ease of use, compatibility, intention to use); each question includes a 7-point Likert scale, from 1 (worst) to 7 (best). The scoring is calculated for each section and is given by the average of the responses in that section, ranging from 1 (worst) to 7 (best).
Questionnaire for satisfaction | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  This is an ad-hoc questionnaire designed to measure satisfaction with healthcare services. Each question uses a 5-point Likert scale, ranging from 1 (unsatisfied) to 5 (very satisfied).
System Usability Scale - SUS | Within 7 days after the end of the 6-week observation/rehabilitation period
  The SUS is a 10 items questionnaire evaluating the perceived usability of a technological system or device. Each item is scored on a Likert scale from 0 to 5, and the total score range from 0 to 100. Higher scores are indicative of higher perceived usability.
Questionnaire for costs | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  Ad-hoc questionnaire to evaluate the costs (direct healthcare costs, direct non-healthcare costs, indirect costs) incurred by the patient, in euros.
Questionnaire for perception of problems and solution complexity | Baseline; within 7 days after the end of the 6-week observation/rehabilitation period
  It is an ad-hoc questionnaire for perception of problems and solution complexity. Each question utilizes a 5-point Likert scale, ranging from 1 (low complexity) to 5 (very complex).
Incremental cost-utility ratio | During the study, an average of 14 months
  The incremental cost-utility ratio (ICUR) will serve as the key metric of the Cost-utility analysis, and it is calculated as the ratio between differences in costs and differences in utility across the analysis groups. Cost-utility analysis will assess and compare the efficiency of alternative rehabilitation interventions by measuring health outcomes in terms of utility, a measure of general well-being or quality of life (subjective measures), relative to the costs incurred to achieve these outcomes. Utilities will be evaluated using standardized measures based on quality of life. Each health condition identified through generic health-related quality of life questionnaires (EQ-5D-DL) will be associated with available utility scores specific to Italy.
Incremental cost-effectiveness ratio | During the study, an average of 14 months
  The incremental cost-effectiveness ratio (ICER) is calculated by dividing the difference in costs between the alternative rehabilitation models tested in the clinical study by the difference in clinical outcomes (physical units - objective measures). It will be used as the key metric of the cost-effectiveness analysis, that will compare the costs and clinical outcomes of the alternative rehabilitation models being studied. The ICER represents the additional cost incurred to achieve an incremental unit of effectiveness, that will be assessed considering primary and secondary outcomes.
Financial impact (differences in direct health costs) | During the study, an average of 14 months
  From the perspective of the payer, the expected outcome of the budget impact analysis is the assessment of the financial impact (differences in direct health costs) over a 3-5 year period for the diffusion of a mix of robotic-based rehabilitations, compared to conventional rehabilitation or a robotic solution. The financial impact will be assessed by considering the direct health costs associated with the different rehabilitation regimes, varying projections of robotic market uptake, and the degrees of substitutability between the compared rehabilitation regimes.
Working-Related Quality of Life | During the study, an average of 14 months
  The Work-Related Quality of Life (WRQoL) scale is a 23-item psychometric instrument designed to measure employees' perceived quality of working life across six psychosocial sub-factors. In this context, the WRQoL scale will be administered to healthcare professionals to assess and better understand their work-related quality of life. Each response will be rated on a 5-point scale (1 to 5).

CONTACTS AND LOCATIONS:
Overall Officials: Irene G Aprile, MD, PhD, Study Director — IRCCS Fondazione Don Carlo Gnocchi; Christian Lunetta, Principal Investigator — IRCCS Istituti Clinici Scientifici Maugeri; Roberto De Icco, Principal Investigator — IRCCS Fondazione Mondino; Carlo Trompetto, Principal Investigator — IRCCS Ospedale Policlinico San Martino; Ennio Ferlazzo, Principal Investigator — COT Istituto Clinico Polispecialistico; Silvana Quaglini, Principal Investigator — Università di Pavia; Giuseppe Turchetti, Principal Investigator — Università Sant'Anna di Pisa; Leandro Pecchia, Principal Investigator — Campus Bio-Medico University
Locations (13):
- Italy (13):
  - Fondazione Don Carlo Gnocchi, Centro Gala, Acerenza
  - IRCCS Istituti Clinici Scientifici Maugeri, Bari
  - IRCCS Ospedale Policlinico San Martino, Genova
  - COT, Cure Ortopediche Traumatologiche, Istituto Clinico Polispecialistico, Messina
  - Fondazione Don Carlo Gnocchi, IRCCS Santa Maria Nascente, Milan
  - IRCCS Istituti Clinici Scientifici Maugeri, Milan
  - IRCCS Istituti Clinici Scientifici Maugeri, Montescano
  - IRCCS Fondazione Mondino, Pavia
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria della Provvidenza, Rome
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria al Mare, Salerno
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Sant'Angelo dei Lombardi
  - IRCCS Istituti Clinici Scientifici Maugeri, Telese Terme
  - Fondazione Don Carlo Gnocchi, Polo specialistico riabilitativo, Tricarico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the publication will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning six months after the publication, with no end date.
Access Criteria: Access will be provided to the general scientific community and any interested researchers, for any type of analysis or secondary research use. The data will be made available on a public data-sharing platform such as Zenodo, or Figshare.